CLINICAL TRIAL: NCT06195280
Title: Prospective, Multicenter Study Evaluating the Diagnostic Performance of the 3DT1 Sequence in Magnetic Resonance Imaging for Superficial Endometriosis
Brief Title: SUPerficial ENDometriosis In Magnetic Resonance Imaging
Acronym: SUPENDIM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients were included in this study.
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A01336-39
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Magnetic Resonance Spectroscopy; Laparoscopy

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- superficial endometriosis (Experimental): Endometriosis is a chronic, estrogen-dependent inflammatory disease secondary to tissue growth outside the uterine cavity, affecting approximately 10% of women of childbearing age.
  Interventions: Radiation: Magnetic resonance imaging, 3DT1 sequence; Procedure: Laparoscopy

INTERVENTIONS:
Radiation: Magnetic resonance imaging, 3DT1 sequence — The patient will have an exploration pelvic Magnetic Resonance Imaging lasting approximately 15 to 20 minutes, without systematic injection of contrast product.
Procedure: Laparoscopy — After Magnetic Resonance Imaging, the patient will benefit from a laparoscopy under general anesthesia lasting an average of one hour.

SUMMARY:
The purpose of the study is to determine the correlation between the diagnosis of Superficial endometriosis by the 3DT1 sequence on Magnetic resonance imaging and the histology obtained by laparoscopy.

DETAILED DESCRIPTION:
This is a prospective, multicenter, non-randomized study evaluating the diagnostic performance of Magnetic Resonance Imaging in superficial endometriosis.

The duration of the patient's participation in the study is a maximum of 15 months depending on the length of the screening period and the time between Magnetic Resonance Imaging and laparoscopy.

After selection, the investigator will check the patient's eligibility and offer her the study. If she accepts and signs the informed consent form, the patient will have an exploratory pelvic Magnetic Resonance Imaging lasting approximately 15 to 20 minutes, without systematic injection of contrast product.

After Magnetic Resonance Imaging, the patient will benefit from a laparoscopy under general anesthesia lasting an average of one hour.

ELIGIBILITY:
Inclusion Criteria :

* Age ≥ 18 years;
* Non-menopausal patient;
* Patient scheduled for exploratory laparoscopy;
* Patient requiring a preoperative pelvic MRI
* Patient having been informed and having signed an informed consent form.

Exclusion Criteria :

* Classic contraindications to magnetic resonance imaging;
* Contraindications to anesthesia for exploratory laparoscopy;
* Contraindication to surgery following the findings of magnetic resonance imaging results;
* Patient with endometrioma > 4 cm;
* Patient with known deep endometriosis;
* Patient uncooperative with protocol requirements or unable to attend the center for scheduled visits;
* Pregnant woman or woman of childbearing age, without effective contraception or breastfeeding;
* Patient participating in another clinical trial, or during a period of exclusion from another clinical trial;
* Patient under guardianship, under curatorship or subject to legal protection, persons deprived of liberty by a judicial or administrative decision, persons subject to psychiatric care and admitted to a health or social establishment;
* Patient not beneficiary of a social security system
* Patient under State Medical Aid.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Endometriosis is a chronic, estrogen-dependent inflammatory disease secondary to tissue growth outside the uterine cavity, affecting approximately 10% of women of childbearing age.
Enrollment: 0 (Actual)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Correlation between the diagnosis of superficial endometriosis by the 3DT1 sequence in Magnetic Resonance Imaging and the histology obtained by laparoscopy | between 30 and 150 days
  The diagnostic validity of Magnetic resonance imaging compared to laparoscopy will be determined by correlation between the locations of the sites screened on Magnetic resonance imaging (Douglas cul de sac, vesicouterine cul de sac, right ovarian fossa, left ovarian fossa, right broad ligament, left broad ligament) and histologically confirmed endometriotic implants at these sites.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Blomet, Paris, France